CLINICAL TRIAL: NCT03485716
Title: Metabolic Dynamics During Physical Activity Under Normobaric Normoxia or Moderate Hypoxia - a Pilot Study
Brief Title: Metabolic Dynamics During Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Michael Boschmann, Dr. Michael Boschmann, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Hypoxitrain 2
Record Dates: First submitted 2018-03-19; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Healthy Men and Women
Keywords: metabolism; metabolome; physical activity; hypoxia
MeSH Terms: conditions — Motor Activity; Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- running under hypoxia - first (Experimental): running under hypoxia (first day) and normoxia (second day)
  Interventions: Other: running on a treadmill under normoxia or hypoxia
- running under normoxia - first (Active Comparator): running under normoxia (first day) and hypoxia (second day)
  Interventions: Other: running on a treadmill under normoxia or hypoxia

INTERVENTIONS:
Other: running on a treadmill under normoxia or hypoxia — * 30 min running (60% VO2max) on a treadmill under hypoxia (O2: 14%)
  * 30 min running (60% VO2max) on a treadmill under normoxia (O2: 20%)

SUMMARY:
The aim of this study is to systematically Analyse the metabolome in capillary blood of healthy men and women at rest and during defined standardized physical activity under normobaric normoxia or hypoxia with a specific focus on metabolites and metabolic pattern related to energy metabolism. The metabolome analyses in capillary blood could give us also or more detailed insight into erythrocyte metabolic physiology because it is known for a longer time that the primary metabolism of the erythrocyte reflects its Oxygen Saturation via the glycolytic metabolites / intermediates pattern.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* written informed consent

Exclusion Criteria:

* known cardio-vascular, lung, metabolic, endocrine, hematologic, kidney or neurologic diseases
* pregnancy, lactating period
* unability to understand study content and aims and to give written informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in capillary lactate/pyruvate Ratio (dimension-free) | t = 0 min (before exercise); t = 10, 20 and 30 min during exercise; t = 50 and 60 min during recovery
  marker for the ratio between anaerobic / aerobic glycolysis

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boschmann, Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charite University Medicine, ECRC, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No